CLINICAL TRIAL: NCT00144443
Title: Kansas City Community Environmental Remediation And Training (KC CERT)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not completed
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: US Department of Housing and Urban Development (U.S. Federal Agency); The healthy Homes Network of Kansas City, Missouri (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RG00002078; GL01.3714
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Asthma; Rhinitis; Allergy
Keywords: Aerobiology; Asthma; Indoor Fungi; Allergen; Home Remediation
MeSH Terms: conditions — Asthma; Rhinitis; Hypersensitivity

INTERVENTIONS:
Behavioral: Basic home repair
Behavioral: Asthma Trigger Education

SUMMARY:
Objective: Our overall objective is to test the hypothesis that the health of children with chronic respiratory symptoms or chronic exposures to environmental hazards can be improved through a combination of standard home maintenance interventions and a set of interim controls and targeted repair interventions.

I. Background:

The Bi-State Kansas City Enhanced Enterprise Community (KCEEC) is one of pervasive poverty, unemployment and general distress. This same area is also an area of poor environmental health with a disproportionate number of children with lead poisoning, asthma, and home injuries.

In May 2001, the Metropolitan (Kansas City) Health Council released a report urging the implementation of strategies to address this growing concern. They stated, "Environmental assessments and interventions in homes, schools, and workplaces are needed to promote indoor air quality and thereby help prevent asthma and asthma flare-ups," in combination with the need for, "trained community-based peer educators needed to work with families/communities in areas of high asthma incidence,". The need for major rehabilitation is echoed in the 1999 Consolidated Plan, as well as by most community development and housing officials.

The KC CERT project responds to these concerns by demonstrating low-cost, replicable intervention strategies that can have an impact on the health and safety of children and their families. By providing training and employment opportunities to residents in high-risk areas to assess, prevent and remediate environmental hazards, this project promotes sustained systematic change within the KCEEC.

DETAILED DESCRIPTION:
This study is an observational study. It will be managed by a project director for HHN and the Environmental Health Program Manager for CMH. Following enrollment in the study, a health assessment focusing on specific respiratory problems and lead exposure will be performed. Eligible subjects must be between the ages of 2 and 17 years of age, and stay in the home a minimum of 4 nights per week.

The home environment will also be assessed using a specific set of on-site and laboratory sampling and analyses. Once study analyses are complete, a report will be written and provided to the family. The health and home assessments will be used in the presentation of in-home education related to specific strategies for creating and maintaining a safe and healthy home. Once the initial assessments are complete, the family will receive a set of standard and targeted interventions that together total no more than $2000 in value. If the house is in need of more than $2000 worth of interventions, the family would not qualify to participate in this study and would be offered alternative resources through the HHN, and the UMKC Center for the City, Home Center.

The interim controls recommended in the assessment will be provided within 60 days of the in-home education. These interim controls include a set of standard interventions that will be provided in all homes and, in addition, a set of site-specific or targeted interventions based on the assessment findings. Six months after the interventions have been implemented, the child's health and the home will be assessed using the same instruments, procedures, questionnaires, and the same number and type of samples as in the initial assessment will be taken. This will ensure consistency and quality in data gathering.

Recruitment of Subjects:

The Healthy Homes Network will recruit participants from community physicians and clinics, and organizations affiliated with the HHN including health departments and housing authorities, the CMH Emergency Room, the CMH Allergy Clinic, other CMH primary care clinics. HHN will recruit through advertising in the media if necessary (see proposed ad included), but the CMH name or LOGO will not appear in the ad. Subjects will be referred to CMH for health evaluations.

Expected Sample Size: Total study: 200 CMH only: 200

Inclusion Criteria:

Participants that qualify for the study will have one of the following health conditions: persistent asthma as defined by NHLBI guidelines, chronic respiratory symptoms, and/or have lead levels equal to or above 15 micrograms per deciliter. They must be between the ages of 2 and 17 years of age, and stay in the home a minimum of 4 nights per week and, they should reside in the KCEEC (Defined as the city limits of Kansas City Kansas or Kansas City Missouri). They will also have lived in the same housing, either rental or self-owned, for at least 6 months and have a reasonable expectation of remaining in this housing for at least one additional year.

To qualify for the intervention phase of the study done by HHN, the home must have no more than $2000 estimated intervention costs. Examples of houses that would not qualify include: A house that needs a new roof, a house with extensive amounts of flaking lead paint, a house with significant structural problems.

Exclusion Criteria:

Any children who do not meet the age and residency requirements. Any home with more than $2000 worth of maintenance and repair problems. Any home with emergent, life threatening conditions. Children with other chronic diseases (leukemia, diabetes etc) will be referred through the HHN and CMH to appropriate medical services, agencies, organizations and other community resources.

There is only one study group (the immediate intervention group). In this group, the child's health will be evaluated, the home environmental health will be assessed and reported to the family, and the family will receive in-home education. Within 60 days of the in-home education, a series of interim controls for the home will be provided by HHN using a specific set of standard interventions and a site-specific set of targeted interventions based on the assessment findings. The home will be checked to ensure the interventions were properly done. After 6 months, the child's health will be reevaluated and the environmental health of the home will be assessed a second time to evaluate the impact on the child's health.

Observations/Measurements:

Goal 1: Demonstrate improvement in overall health and chronic symptoms in children

Pre/Post Measures:

1. Health Assessment Questionnaire
2. Asthma severity (assigned by blinded physician - based on health assessment and spirometry [for children >5 years old] )
3. Medication dosage (taken from family health information)
4. Blood lead level (measured in clinical lab)
5. Allergen Specific IgG & IgE (measured in clinical lab)
6. Number of days of school missed (taken from family health survey)
7. Number of days as in-patient in hospital (taken from hospital records)
8. Number of visits to physician/ER (taken from clinic records)
9. Quality of life rating (from SF12 form)
10. Asthma specific quality of life rating (Juniper et. al.)

Goal 2: Reduce specific environmental hazards potentially affecting health through interventions

Pre/Post Measures:

1. IAQ Survey (On-site analyses for Temp. RH. CO2, CO, THC, VOC, TVOC)
2. Allergen content in house dust (lab measurement by immunoassay)
3. Total Particulate Analysis (on-site laser particle analysis)
4. Airborne spore levels (measured by spore trap determination)
5. Chemical Exposure Hazard (home assessment and site-specific chemical analysis)

Goal 3: Demonstrate effectiveness of low-cost intervention

Measures:

a. Differential in environmental exposure factors and health symptom factors before enrolment in study and 6 months after home interventions. (Evaluated by statistical methods; mostly students t-test). Power analysis indicates adequate power to detect a 50% change in allergen level in dust at a 95% confidence level with 66 houses in each group.

Goal 4: Reduce specific environmental hazards potentially affecting health through in-home education.

Pre/Post Measures:

1. IAQ Survey (On-site analyses for Temp. RH. CO2, CO, THC, TVOC, O3)
2. Allergen content in house dust (lab measurement by immunoassay)
3. Total Particulate Analysis (on-site laser particle analysis)
4. Airborne spore levels (measured by spore trap determination)
5. Chemical Exposure Hazard (home assessment and site-specific chemical analysis)

ELIGIBILITY:
Inclusion Criteria:

Participants that qualify for the study will have one of the following health conditions:

* Persistent asthma as defined by NHLBI guidelines
* Chronic respiratory symptoms,
* And/or have lead levels equal to or above 15 micrograms per deciliter.
* They must be between the ages of 2 and 17 years of age
* Stay in the home a minimum of 4 nights per week
* They should reside in the KCEEC (Defined as the city limits of Kansas City Kansas or Kansas City Missouri).
* They will also have lived in the same housing, either rental or self-owned, for at least 6 months and have a reasonable expectation of remaining in this housing for at least one additional year.

To qualify for the intervention phase of the study done by HHN,

* The home must have no more than $2000 estimated intervention costs. Examples of houses that would not qualify include: A house that needs a new roof, a house with extensive amounts of flaking lead paint, a house with significant structural problems.

Exclusion Criteria:

* Any children who do not meet the age and residency requirements.
* Any home with more than $2000 worth of maintenance and repair problems. - Any home with emergent, life threatening conditions.
* Children with other chronic diseases (leukemia, diabetes etc) will be referred through the HHN and CMH to appropriate medical services, agencies, organizations and other community resources.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200
Dates: Start 2003-03; Study Completion 2005-05

PRIMARY OUTCOMES:
Reduction in home airborne fungal spore levels.
Reduction in home allergen exposure.

SECONDARY OUTCOMES:
Reduction in healthy care utilization
Improvement in quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Charles S Barnes, Ph.D., Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

REFERENCES:
- [Background] Portnoy JM, Kwak K, Dowling P, VanOsdol T, Barnes C. Health effects of indoor fungi. Ann Allergy Asthma Immunol. 2005 Mar;94(3):313-9; quiz 319-22, 390. doi: 10.1016/S1081-1206(10)60982-9. PMID 15801241